CLINICAL TRIAL: NCT00142805
Title: Safety, Tolerability and Efficacy Study of Tricaprilin (AC-1202) Administered for Ninety Days in Subjects With Probable Alzheimer's Disease of Mild to Moderate Severity
Brief Title: Tricaprilin in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KET-04-001
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer's Disease
Keywords: ketones; Apolipoprotein E; ApoE genotype; cognitive function; glucose metabolism
MeSH Terms: conditions — Alzheimer Disease; Ketosis | interventions — tricaprylin; AC-1202

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AC-1202 (Active Comparator): Tricaprilin formulation, once daily. Administered orally
  Interventions: Drug: Tricaprilin
- Matching Placebo to AC-1202 (Placebo Comparator): Placebo formulation, once daily. Administered orally
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tricaprilin — Powder formulation will be mixed in a liquid (approximately 8 oz).
  Other Names: AC-1202
  Arms: AC-1202
Other: Placebo — Powder formulation will be mixed in a liquid (approximately 8 oz).
  Other Names: Matching placebo to AC-1202
  Arms: Matching Placebo to AC-1202

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and effectiveness of tricaprilin administered once a day for ninety days in subjects with mild to moderate, probable Alzheimer's disease.

DETAILED DESCRIPTION:
Substantial scientific evidence has shown that defects in glucose metabolism occur in Alzheimer's disease. Attempts to compensate for the reduced cerebral metabolic rates in AD have met with some success. Treatment of AD patients with high doses of glucose and insulin will raise cognitive scores. However, this effect is slight, and high doses of insulin can have adverse consequences. Administration of ketone bodies or their metabolic precursors such as medium chain triglycerides (MCTs) presents an attractive alternative to glucose and insulin. In a preliminary study, tricaprilin, an MCT, demonstrated pharmacological activity and statistically significant efficacy in improving short-term memory and attention performance after a single dose.

Participants will be randomized to receive either tricaprilin or a matching placebo, administered once a day by mixing powder in a glass of liquid. The treatment period will last 90 days, followed by a 2-week washout period. Each patient will be seen 5 times: at screening, baseline, and post-baseline days 45, 90, and 104. The visits will include physical and/or neuropsychological examinations, electrocardiograms (ECGs) and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form signed by patient and caregiver
* Diagnosis of probably Alzheimer's disease of mild to moderate severity
* Age 50 or older
* If female, 2 years postmenopausal or surgically sterile
* Hearing, vision, and physical abilities adequate to perform assessments (corrective aids allowed)
* Caregiver to attend all visits, perform assessments, and supervise administration of study medication
* CT or MRI within 24 months prior to screening compatible with a diagnosis of probably Alzheimer's disease
* Modified Hachinski Ischemia Scale score of 4 or less
* ADAS-Cog score between 15 and 35 inclusive at screening
* MMSE score between 14 and 24 inclusive at screening
* Stable medical condition for 3 consecutive months immediately prior to baseline
* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Any condition that would, in the opinion of the Principal Investigator, render the patient or the caregiver unsuitable for the study, or place them at substantial risk of adverse outcome
* Unwillingness or inability of the patient and/or caregiver to fulfill the requirements of the study
* Resident in a skilled nursing facility
* Any significant neurological disease other than probable AD (e.g. Parkinson's disease, Huntington's disease, brain tumor, normal pressure hydrocephalus, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of stroke, or history of head injury requiring hospitalization)
* An alternate cause for dementia other than AD as determined by a required CT or MRI scan within 24 months prior to screening
* Current history of major psychiatric disorder
* Major depression as determined by a Cornell Scale for Depression in Dementia
* Clinically significant hypothyroidism
* Clinically significant B12 deficiency
* Unstable or clinically significant cardiovascular disease
* Diabetes of any type
* History of tertiary syphilis
* Cancer within 3 years prior to baseline, with the exception of squamous and basal cell carcinoma
* Vital sign abnormalities
* Clinically significant renal disease or insufficiency
* Clinically significant hepatic disease or insufficiency
* Alcohol consumption greater than 2 oz of spirits per day or 14 oz per week (1 oz of spirits is equal to 6 oz of wine or 12 oz of beer)
* Current history of alcohol abuse or other substance abuse within 24 months prior to baseline
* Known HIV infection
* Use of any investigational compound within 30 days prior to screening
* Use of prohibited medications (contact site for details)
* Prior or current use of medium-chain triglycerides (MCTs) for medical purposes
* Known allergies to coconut oil

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2004-11-04 (Actual); Primary Completion 2006-06-29 (Actual); Study Completion 2007-01-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment related adverse events | 104 days
  AE incidence rate per treatment group

SECONDARY OUTCOMES:
Pharmacokinetics (PK) profile of tricaprilin | Baseline, Day 45, Day 90
  Correlations between the Cmax serum BHB level on Day 90 and the change from baseline total score for the three efficacy scales was determined by the Pearson correlation statistics
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | 90 days
  Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog 11) is an 11- item cognitive subscale that objectively measures memory, language, orientation, and praxis with a total score range of 0 (no impairment) to 70 (severe impairment)
Clinical Global Impression of Change | 90 days
  Clinician's global impression rated with Alzheimer's Disease cooperative Study - Clinical Global Impression of Change (ADCS-CGIC). The rating is from marked improvement to marked worsening.
Mini-Mental State Exam (MMSE) | 90 days
  Change in MMSE

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - 21st Century Neurology, a division of Xenoscience Inc., Phoenix, Arizona
  - Comprehensive NeuroScience, Cerritos, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pharmacology Research Institute, Northridge, California
  - The Southwest Institute for Clinical Research, Rancho Mirage, California
  - Pharmacology Research Institute, Riverside, California
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Florida
  - Meridien Research, Brooksville, Florida
  - Baumel-Eisner Neuromedical Institute, Inc., Fort Lauderdale, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Comprehensive NeuroScience, Melbourne, Florida
  - Baumel-Eisner Neuromedical Institute, Miami Beach, Florida
  - Anchor Research Center, Naples, Florida
  - Renstar Medical Research, Ocala, Florida
  - Comprehensive NeuroScience, St. Petersburg, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Radiant Research, Chicago, Illinois
  - Multi-Specialty Research Associates of North Carolina, Raleigh, North Carolina
  - Radiant Research, Portland, Oregon
  - Radiant Research, Dallas, Texas
  - Research Across America, Dallas, Texas
  - Radiant Research, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas

REFERENCES:
- [Background] Blass JP, Zemcov A. Alzheimer's disease. A metabolic systems degeneration? Neurochem Pathol. 1984 Summer;2(2):103-14. doi: 10.1007/BF02834249. PMID 6544385
- [Background] Reiman EM, Caselli RJ, Yun LS, Chen K, Bandy D, Minoshima S, Thibodeau SN, Osborne D. Preclinical evidence of Alzheimer's disease in persons homozygous for the epsilon 4 allele for apolipoprotein E. N Engl J Med. 1996 Mar 21;334(12):752-8. doi: 10.1056/NEJM199603213341202. PMID 8592548
- [Background] Small GW, Ercoli LM, Silverman DH, Huang SC, Komo S, Bookheimer SY, Lavretsky H, Miller K, Siddarth P, Rasgon NL, Mazziotta JC, Saxena S, Wu HM, Mega MS, Cummings JL, Saunders AM, Pericak-Vance MA, Roses AD, Barrio JR, Phelps ME. Cerebral metabolic and cognitive decline in persons at genetic risk for Alzheimer's disease. Proc Natl Acad Sci U S A. 2000 May 23;97(11):6037-42. doi: 10.1073/pnas.090106797. PMID 10811879
- [Background] Swaab DF, Lucassen PJ, Salehi A, Scherder EJ, van Someren EJ, Verwer RW. Reduced neuronal activity and reactivation in Alzheimer's disease. Prog Brain Res. 1998;117:343-77. doi: 10.1016/s0079-6123(08)64027-3. PMID 9932420
- [Background] Laffel L. Ketone bodies: a review of physiology, pathophysiology and application of monitoring to diabetes. Diabetes Metab Res Rev. 1999 Nov-Dec;15(6):412-26. doi: 10.1002/(sici)1520-7560(199911/12)15:63.0.co;2-8. PMID 10634967
- [Background] Kashiwaya Y, Takeshima T, Mori N, Nakashima K, Clarke K, Veech RL. D-beta-hydroxybutyrate protects neurons in models of Alzheimer's and Parkinson's disease. Proc Natl Acad Sci U S A. 2000 May 9;97(10):5440-4. doi: 10.1073/pnas.97.10.5440. PMID 10805800
- [Derived] Henderson ST, Poirier J. Pharmacogenetic analysis of the effects of polymorphisms in APOE, IDE and IL1B on a ketone body based therapeutic on cognition in mild to moderate Alzheimer's disease; a randomized, double-blind, placebo-controlled study. BMC Med Genet. 2011 Oct 12;12:137. doi: 10.1186/1471-2350-12-137. PMID 21992747
- [Derived] Henderson ST, Vogel JL, Barr LJ, Garvin F, Jones JJ, Costantini LC. Study of the ketogenic agent AC-1202 in mild to moderate Alzheimer's disease: a randomized, double-blind, placebo-controlled, multicenter trial. Nutr Metab (Lond). 2009 Aug 10;6:31. doi: 10.1186/1743-7075-6-31. PMID 19664276
- See also: Accera Pharmaceuticals Clinical Trials Query Form — http://www.accerapharma.com/